CLINICAL TRIAL: NCT05073237
Title: Effects of Novel Estrogens on Glucose and Lipids in Postmenopausal Prediabetic Women Veterans
Acronym: CE/BZA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENDA-009-20F; 1IK2CX002225-01A1 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Menopause; Prediabetes; Obesity
Keywords: Menopause; prediabetes; diabetes; obesity; hot flushes; hormones; estrogen; bazedoxifene
MeSH Terms: conditions — Prediabetic State; Obesity; Diabetes Mellitus; Hot Flashes | interventions — Estrogens, Conjugated (USP); bazedoxifene

STUDY DESIGN:
Intervention Model Description: In the current study, 40 women veterans with obesity, prediabetes and menopause who are experiencing bothersome menopause symptoms will be enrolled and randomized to receive either 16 weeks of CE/BZA or 16 weeks of placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double blind, placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conjugated estrogens/bazedoxifene (CE/BZA) (Experimental): Participants assigned to CE/BZA will receive a daily tablet containing conjugated estrogens 0.45 mg and bazedoxifene 20 mg. Recommended and only FDA approved dosage is one CE/BZA tablet daily, taken without regard to meals. Tablets should be swallowed whole. If a dose of BZA/CE is missed, participants will be instructed to take it as soon as remembered unless it is almost time for the next scheduled dose. They should not take two doses at the same time. The dose is one tablet per day independent of weight and fat mass. Participants will be provided with information about BZA/CE and its potential side effects and contraindications.
  Interventions: Drug: conjugated estrogens/bazedoxifene (CE/BZA)
- Placebo (Placebo Comparator): Participants assigned to placebo will receive a daily tablet. To assure the blind is maintain, participants in the placebo group will be given the same instructions for taking the study medication. Tablets should be swallowed whole. If a dose, participants will be instructed to take it as soon as remembered unless it is almost time for the next scheduled dose. They should not take two doses at the same time. The dose is one tablet per day independent of weight and fat mass. Participants will be provided with information about CE/BZA and its potential side effects and contraindications, again to maintain the blind.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Daily placebo tablet
  Arms: Placebo
Drug: conjugated estrogens/bazedoxifene (CE/BZA) — Participants assigned to CE/BZA will receive a daily tablet containing conjugated estrogens 0.45 mg and bazedoxifene 20mg.
  Other Names: DUAVEE
  Arms: conjugated estrogens/bazedoxifene (CE/BZA)

SUMMARY:
The purpose of this study is to determine the effect of a novel menopause hormone therapy on blood sugar (glucose) and blood and liver fats (lipids) in obese menopausal women Veterans.

DETAILED DESCRIPTION:
Menopause is a natural process characterized by estrogen deficiency that results in several undesirable metabolic changes, including increase in body fat, decrease in lipid oxidation, impairment in glucose tolerance, and hyperinsulinemia. One in four women dies of cardiovascular disease (CVD), and with the increase in life expectancy, many women will spend almost half of their lives in a postmenopausal state of estrogen deficiency that predisposes them to metabolic syndrome, hyperlipidemia (HLD) and type 2 diabetes (T2D) resulting in overall increased risk for CVD. Menopausal hormone therapy (MHT) is beneficial if administered in early menopausal women, age 50-60 years . The most promising and novel MHT involves the combination of conjugated estrogens (CE) with the selective estrogen receptor modulator bazedoxifene (BZA) in a single tablet. The major innovation of CE/BZA is that it provides all the advantages of CE treatment without the use and side effects of a progestin. Moreover, an important beneficial effect of estrogen is also to prevent postmenopausal metabolic disorders . One of the most comprehensive research initiatives undertaken on the postmenopausal health of women, The Women's Health Initiative (WHI), involved nearly 4,000 women Veterans. The studies from WHI show how military service affects women's longevity and overall health as compared to non-Veterans. The data from WHI shows that women Veterans have higher all-cause mortality rates than non-Veterans and higher hip fracture rates despite similar risk factors. Also, women Veterans <65 years at WHI enrollment were more likely to have experienced prior hysterectomy and early hysterectomy before age 40 compared with non-Veterans.

Additionally, information about the effectiveness of CE/BZA as MHT in women with abnormal glucose is lacking. In that regard, there is a critical need to determine the effects of CE/BZA on beta cell function in obese menopausal women with early glucose abnormalities, primarily in the pre-diabetes and early diabetes stages, and prevent evolution toward full-blown diabetes as these women are at higher risk for CVD.

In the current study, 40 women Veterans with obesity, prediabetes and menopause who are experiencing bothersome menopause symptoms will be enrolled and randomized to receive either 16 weeks of CE/BZA or 16 weeks of placebo to find the effect of the drug on glucose and lipids metabolism.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women veterans within 5 years of menopause.

Menopause is defined as:

* women with intact uterus and last menstrual period >1 year ago but <5 years ago
* Age 50-60 years
* BMI 27-34.9kg/m2 (Overweight and low risk Class 1 Obesity)
* Symptomatic (moderate to severe vasomotor symptoms)
* Fasting glucose 100-150mg/dl or/or HbA1c >5.7%- and <7% (two abnormal test can be fasting glucose or HbA1c or combination of the two in the past 6 months).
* Triglycerides < 200 mg/dl
* GFR >60mL/min
* Normal mammogram within the past 12 months

Exclusion Criteria:

* Amenorrhea from other causes (Hyperandrogenemia and anovulation)
* Recent weight change (>10 lbs in the last 3 months), intended or unintended
* Vulnerable populations (employees, students, individuals with impaired decision making capacity, pregnant women, prisoners, terminally ill, and children)
* Change in lipid lowering agent in the last 3 months
* Use of glucose lowering agents in the last 3 months
* Concurrent conditions including HIV, uncontrolled hyperthyroidism, uncontrolled hypothyroidism or less than 3 months since addition or change in thyroid hormone modulating medications, current use of drugs known to promote significant weight changes, menopause hormone therapy use within 3 months
* Contraindications to estrogens (history of thromboembolic disorder, coronary artery or cerebrovascular disease, clotting disorders (Antiphospholipid antibody syndrome, protein C deficiency, protein S deficiency, AT III deficiency, factor V leiden), severe liver disease, history of breast or uterine cancer or unexplained vaginal bleeding)
* Plan for major surgery or prolonged immobilization within 6 month period
* MRI Absolute contraindications

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
change in beta cell function | Change in beta cell function between baseline and 16 weeks
  beta cell function will be evaluated via oral glucose tolerance test at baseline and after 16 weeks of treatment.

SECONDARY OUTCOMES:
change in liver fat | Change in Liver fat between baseline and 16 weeks
  Change in liver fat will be evaluated via MRI-PDFF between baseline and after 16 weeks of treatment.
change in serum lipidomics | Change in serum lipidomics between baseline and 16 weeks
  Change in serum lipidomics will be evaluated via UPLC-MS/MS at baseline and after 16 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Lovre, MD, Principal Investigator — Southeast Louisiana Veterans Health Care System, New Orleans, LA
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No